CLINICAL TRIAL: NCT03339271
Title: Technology-enhanced Transitional Palliative Care for Family Caregivers in Rural Settings
Brief Title: Technology-enhanced Transitional Palliative Care for Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Joan M. Griffin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-005188; R01NR016433 (NIH)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-Enhanced Group (Active Comparator): Family caregivers will have daily visits from the study nurse while the patient is in the hospital and will receive weekly technology-enhanced support (video chats) from the study nurse for 8 weeks after the patient is discharged from the hospital.
  Interventions: Behavioral: Technology-Enhanced Support
- Usual Care Group (Active Comparator): Family caregivers will have usual care support from the doctors and nurses to plan for taking care of the patient upon return home and will receive a weekly telephone call for 8 weeks after the patient is discharged from the hospital.
  Interventions: Behavioral: Usual Care Support

INTERVENTIONS:
Behavioral: Technology-Enhanced Support — The study nurse will meet with the caregiver daily until patient is discharged from the hospital. The caregiver will take home an iPad upon discharge, and will have an initial video chat with the study nurse within 24-48 hours of hospital discharge and weekly for 8 weeks after that.
  Arms: Technology-Enhanced Group
Behavioral: Usual Care Support — The patient's doctor and nurses with input from the Palliative Care service will help the caregiver make a plan for discharge of the patient, and for taking care of the patient upon discharge. Someone from the study team will call the caregiver once a month for the duration of the study after the patient discharges from the hospital.
  Arms: Usual Care Group

SUMMARY:
The purpose of this study is to evaluate the effect and cost of technology-enhanced transitional palliative care on family caregivers who provide care to a loved one after a hospitalization.

DETAILED DESCRIPTION:
There will be two groups in this randomized control study: technology-enhanced group and usual care group. The total amount of subjects includes both the palliative care recipients and the family caregivers (both the patients and their family caregiver will sign informed consent.)

A family caregiver is broadly defined as the person self-identified as the family member or unpaid friend who is the primary informal caregiver for a patient with a terminal illness. The family caregiver may or may not be a member of the patient's nuclear family.

For the technology-enhanced group, the study nurse experienced in palliative care will have a visit with the caregiver within the first 24 hours after consent, and have daily visits with the caregiver as long as the patient is still in the hospital. During these visits, the nurse will talk to the caregiver about their own self-care needs, begin transitional care planning, and develop Readiness Plans to anticipate care giving needs the caregiver may have when they discharge from the hospital.

For the technology-enhanced group, the caregiver will take an iPad home so that the study team nurse can video chat with them. The iPad will need to be returned upon completion of the study. The study nurse will have a video chat with the caregiver at home within 24-48 hours of discharge from the hospital, and at least weekly for 8 weeks after that. The caregiver and the study nurse may also decide to have other calls on the phone during this time.

For the usual care group, doctors and nurses along with input from the Palliative Care service will help the caregiver make a plan for discharge from the hospital and for taking care of the patient upon discharge. Someone from the study team will call the caregiver once a month to check in for the 6 months after the patient discharges from the hospital.

Both groups will be asked to complete questionnaires before starting the study, and then up to seven more times over the course of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult family caregiver of adult patient hospitalized at Mayo Clinic
* Receives in-hospital palliative care consult
* Family caregiver lives in a Minnesota or Iowa county that is designated as medically under served or rural area

Exclusion Criteria:

* Family caregivers who live in Rochester, Minnesota. (Rochester, Minnesota is not considered a medically under served or rural area.)
* Patients with left ventricular assistive devices, documented chronic pain, use of home infusion pain pumps, or documented addictive behaviors.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane E Holland, PhD, RN, Principal Investigator — Mayo Clinic; Joan M Griffin, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Griffin JM, Holland DE, Vanderboom CE, Kaufman BG, Gustavson AM, Ransom J, Mandrekar J, Dose AM, Ingram C, Fong ZV, Wild E, Weiss ME. Assessing Family Caregiver Readiness for Hospital Discharge of Patients With Serious or Life-Limiting Illness Using Electronic Health Record (EHR) and Self-Reported Data. Health Serv Res. 2025 Jan 28;60(4):e14441. doi: 10.1111/1475-6773.14441. Online ahead of print. PMID 39871699
- [Derived] Kaufman BG, Huang RW, Holland DE, Vanderboom CE, Ingram C, Wild EM, Dose AM, Stiles C, Gustavson AM, Mandrekar J, Van Houtven CH, Griffin JM. Healthcare use and out-of-pocket costs for rural family caregivers and care recipients in a randomized controlled trial. J Am Geriatr Soc. 2024 Aug;72(8):2523-2531. doi: 10.1111/jgs.18934. Epub 2024 May 2. PMID 38698643
- [Derived] Holland DE, Vanderboom CE, Mandrekar J, Borah BJ, Dose AM, Ingram CJ, Griffin JM. A technology-enhanced model of care for transitional palliative care versus attention control for adult family caregivers in rural or medically underserved areas: study protocol for a randomized controlled trial. Trials. 2020 Oct 28;21(1):895. doi: 10.1186/s13063-020-04806-0. PMID 33115524
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Care recipients were not enrolled into this study. All study activities were conducted with the caregivers not the care recipients.
Period: Overall Study
Arm/Group | Technology-Enhanced Group | Usual Care Group
Started | 195 | 189
Completed | 195 | 189
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Family caregivers who live in rural or underserved areas and are caring for a hospitalized patient who has received a palliative care consultation during the hospitalization. Care recipients were not enrolled into this study. All study activities were conducted with the caregivers not the care recipients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Technology-Enhanced Group | Usual Care Group | Total
Number analyzed (Participants) | 195 | 189 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (15.1) | 66.8 (14.3) | 66.7 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 124 | 255
  Male | 64 | 65 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 160 | 123 | 283
  Unknown or Not Reported | 33 | 66 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 167 | 130 | 297
  More than one race | 5 | 10 | 15
  Unknown or Not Reported | 21 | 45 | 66
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 195 | 189 | 384

OUTCOME MEASURES:

1. Primary Outcome: Change in Preparedness for Caregiving Scale Score
Description: The Preparedness for Caregiving Scale captures how well family caregivers feel they are prepared for the multiple aspects of the caregiving role, using a 4-point response set ranging from 0 ("not at all") to 4 ("very well"). A mean score is calculated; higher scores indicate greater preparation for caregiving.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Technology-Enhanced Group: Family caregivers will have in hospital visits from the study nurse while the patient is in the hospital and will receive weekly technology-enhanced support (video chats) from the study nurse for 8 weeks after the patient is discharged from the hospital.
  Technology-Enhanced Support: The study nurse will meet with the caregiver until patient is discharged from the hospital. The caregiver will either use study technology (IPad) or personal technology (personal phone or computer) to have an initial video chat with the study nurse within 24-48 hours of hospital discharge and weekly for 8 weeks after that.
Arm/Group | Technology-Enhanced Group | Usual Care Group
Number analyzed (Participants) | 92 | 72
score on a scale | 0.3 (0.6) | 0.0 (0.7)

2. Secondary Outcome: Change in Communication With Physicians Scale Score
Description: The Communication with Physicians scale will be used to measure the communication skills of the family caregiver. Originally designed for chronic disease self-management behavior, the scale has 3 questions targeting how often the family caregiver prepares a list of questions for the doctor, asks questions, and discusses personal problems across a 6-point response set ranging from "never" to "always." Scores range from 0-5 with higher scores indicating better communication.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Technology-Enhanced Group | Usual Care Group
Number analyzed (Participants) | 92 | 69
score on a scale | 1.0 (1.1) | 0.7 (1.2)

3. Secondary Outcome: Mean Change in Patient Assessment of Chronic Illness Care (PACIC) Score
Description: The mean change in PACIC score. The PACIC was used to obtain family caregiver perceptions of the quality of chronic illness care received by the care recipient. The PACIC is a 20-item caregiver report instrument that measures caregivers' perspectives on the structure of the care for their care recipients and collects caregiver reports on the extent to which their care recipients have received specific clinical services and actions. Each question item is scored on a 5-point scale ranging from 1 to 5 with higher score indicating better care. Total scores range from 0 - 100, lower scores indicate worse care, higher scores indicate better care.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Technology-Enhanced Group | Usual Care Group
Number analyzed (Participants) | 41 | 33
score on a scale | 0.0 (1.0) | -0.1 (0.7)

4. Secondary Outcome: Change in Caregiver Quality of Life Scale - Cancer (CQOL-C) Score
Description: The Caregiver Quality of Life Scale - Cancer (CQOL-C) will be used to measure the family caregiver's quality of life. The CQOL-C is a 35-item self-report measure of the impact on the caregiver's physical, emotional and spiritual well-being and on the relationship with the care recipient. Scores range from 0-140; higher scores indicate worse quality of life.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Technology-Enhanced Group | Usual Care Group
Number analyzed (Participants) | 88 | 69
score on a scale | -7.0 (17.2) | 1.7 (14.3)

5. Secondary Outcome: Mean Change in Bakas Caregiving Outcomes Scale-Revised (BCOS-R) Score
Description: The mean change in BCOS-R score. The Bakas Caregiving Outcomes Scale-Revised (BCOS-R) was used to measure the burden placed on the family caregiver in caring for their loved ones. The BCOS-R contains 16 items that measure changes as indicators of the effect of caregiving on caregivers' lives. The response set uses a 7-point Likert scale that ranges from -3 to -1 = (changed for the worst), 0 = Did not change, +1 to +3 = (changed for the best). Total scores range from -48 to 48, lower scores indicate more negative caregiver outcomes, higher scores indicate more positive caregiver outcomes.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Technology-Enhanced Group | Usual Care Group
Number analyzed (Participants) | 90 | 69
score on a scale | -0.1 (0.5) | -0.1 (0.7)

6. Secondary Outcome: Post Discharge Coping Difficulty Scale (PDCDS) Score
Description: The Post Discharge Coping Difficulty Scale (PDCDS) is a caregiver reported 11-item scale used to measure the degree of difficulty in coping with stress, recovery, self-care and management of medical needs, help and emotional support needed, confidence in self-care and medical management abilities, and adjustment after hospital discharge. The items are measured on an 11-point rating scale that ranges from 0 = Not at all to 10 = extremely, completely, or a great deal. Total scores range from 0 - 110 with lower scores indicating smaller coping difficulty and higher scores indicating greater coping difficulty.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Technology-Enhanced Group | Usual Care Group
Number analyzed (Participants) | 75 | 60
score on a scale | 3.8 (1.9) | 4.1 (1.8)

7. Secondary Outcome: Mean Change in Center for Epidemiological Studies Depression Scale (CESD-10) Score
Description: The mean change in CESD-10 score. The CESD-10 is a caregiver reported 10-item scale used to measure depression. Each question is scored on a 4-point scale, that ranges from 0 = none or rarely to 3 = all of the time. Total scores range from 0- 30, where 0 = no depression and 30 = the most depression.
Time Frame: baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Technology-Enhanced Group | Usual Care Group
Number analyzed (Participants) | 89 | 69
score on a scale | -1.2 (5.8) | 0.4 (5.0)

8. Secondary Outcome: Mean Total Out-of-Pocket Expenditures at 6 Months
Description: The Ambulatory and Home Care Record (AHCR) will be used as the healthcare cost measure. The AHCR is designed to capture costs from a societal perspective, implying that costs from all stakeholders (family care givers, care recipients, and health systems) will be collected.The AHCR captures self-reported utilization and cost information for care provided by all family caregivers and other unpaid caregivers, paid care received at home (e.g., home health care) and outside of the home (e.g., doctor/therapy appointments),as well as medications, supplies, and equipment. Out-of-pocket costs refer to all care-related expenses not paid for by the insurance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Technology-Enhanced Group | Usual Care Group
Number analyzed (Participants) | 151 | 131
dollars
  Health care costs | 571.16 (1008.6) | 503.92 (839.76)
  Food costs | 52.26 (99.76) | 49.26 (93.52)
  Transportation costs | 90.19 (141.51) | 96.98 (144.00)
  Lodging costs | 93.66 (229.56) | 78.5 (215.73)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of the study, approximately 6 months.
Description: Care recipients were not enrolled into this study. All study activities were conducted with the caregivers not the care recipients.
Arm/Group | Technology-Enhanced Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/195 | 0/189
Serious Adverse Events (participants affected / at risk) | 0/195 | 0/189
Other Adverse Events (participants affected / at risk) | 0/195 | 0/189

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03339271/Prot_SAP_000.pdf